CLINICAL TRIAL: NCT07159776
Title: Multiple Digital Biomarkers for Optimization of IBD Care
Acronym: LEGEND-IBD
Status: Not yet recruiting | Type: Observational
Sponsor: Imelda GI Clinical Research Center (Other)
Collaborators: Agentschap Innoveren & Ondernemen (VLAIO) (Unknown)
Responsible Party: Sponsor
Other Study IDs: imelda 202501
Record Dates: First submitted 2025-08-23; First posted 2025-09-08 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Crohn Disease (CD); Ulcerative Colitis (UC); Inflammatory Bowel Disease (IBD)
Keywords: biomarkers; artificial intelligence; wearable; shopping data; life style
MeSH Terms: conditions — Crohn Disease; Colitis, Ulcerative; Inflammatory Bowel Diseases | interventions — Patient Reported Outcome Measures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with IBD: 1. Patients with IBD in longstanding remission (>2 years) (maximum of 20 patients)
  2. Patients with IBD recent event (diagnosis or flare of IBD) (<1year) (minimum 20 patients)
  3. Additional patients with IBD in standard follow up.
  Interventions: Device: monitoring of wearable data, shopping data, biomarkers and patient reported outcomes

INTERVENTIONS:
Device: monitoring of wearable data, shopping data, biomarkers and patient reported outcomes — 1. All participants will receive a wearable device type Corsano Health Cardio watch 287-2 which is provided by the sponsor via Inovigate. Participants will be encouraged to wear the device 24h per day and need to wear the wearable device at least 12 hours per day, preferential during daytime.
  2. All participants will receive a loyalty card (Xtra card Colruyt group) which is provided by the sponsor via Inovigate for food data capturing. The patient is requested to execute all grocery shopping at one of the Colruyt Group stores. He/she will always need to offer the loyalty card to the cashier prior to payment. The purchase receipt will then be automatically sent to the central food data repository at the sponsor set up for this study. Non-food or non-food related data will neither be captured nor stored during the trial.
  3. biomarkers in blood and feaces will be monitored according to standard of care
  4. patient reported outcomes will be monitored according to standard of care

SUMMARY:
To develop digital biomarkers associated with disease activity of inflammatory bowel disease

DETAILED DESCRIPTION:
The trial aims to develop digital biomarkers based on a large dataset of imput data. These data come from diffent sources including wearable data, grocery shopping data, patient reported outcome data, laboratory data and technical exam data. A model will be build that predict disease activity in IBD.

ELIGIBILITY:
Inclusion Criteria:

* Males or females aged > 18 years
* Diagnosis of CD, UC or IBD-unspecified for at least 1 month
* Treatment with conventional or advanced therapy for IBD at initiation of the study
* The patient must have access to an email address
* The patient must be willing to perform all the groceries shopping at any of the Colruyt Group stores during this study, using an Xtra card created by the study team.
* Capacity to independently answer regular digital questionnaires
* Capacity and willingness to use a smartphone and activity tracker

Exclusion Criteria:

* Planned extended (> 1 month) overseas travel during the study period of 12 months, if internet access would be impossible, inconvenient or unaffordable during this time
* Previous colectomy
* Inability to communicate well with investigators or unable to comply with the study requirements
* Significant medical condition interfering with physiological measurements trough a wearable device (heart failure, pacemaker or defibrillator)
* Inclusion or planned inclusion in an interventional IBD-related clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is an open label observational trial with partially blinded data collection (wearable and shopping data blinded for the patient and treating HCP). Patients in the study will not be randomized. Patients will be recruited via planned outpatient visits and day clinic admissions. Patients will be allocated to one of the three target patient groups at the investigator's discretion.
  1. Patients with IBD in longstanding remission (>2 years) (maximum of 20 patients)
  2. Patients with IBD recent event (diagnosis or flare of IBD) (<1year) (minimum 20 patients)
  3. Additional patients with IBD in standard follow up.
  From the moment 60 patients are included, no additional patients can be recruited in group 1 or 3 prior to completion of group 2.
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-09-08 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients in which a flare can be detected based on passive monitoring data. | 1 year

SECONDARY OUTCOMES:
Proportion of patients in which a biomarker flare can be detected based on passive monitoring data | 1 year
Proportion of patients in which an objective disease flare (combination of flare and biomarker flare) can be detected based on passive monitoring | 1 year
Proportion of patients in which a flare can be detected based on food purchase data | 1 year
Proportion of patients in which a biomarker flare can be detected based on food purchase data | 1 year
Proportion of patients in which an objective disease flare (combination of flare and biomarker flare) can be detected based on food purchase data | 1 year

OTHER OUTCOMES:
- Interval between onset of a flare and detection based on passive monitoring data | 1 year
  exploratory outcome
- Subgroup analysis based on the food frequency questionnaire | 1 year
  Exploratory outcome
- Patient satisfaction based on patient experience questionnaire | 1 year
  Exploratory outcome
- Proportion of patients in which (different levels of) disability can be detected based on passive monitoring data | 1 year
  .exploratory outcome
- Proportion of patients in which a change of IBD medication can be detected based on passive monitoring data | 1 year
  Exploratory outcome

CONTACTS AND LOCATIONS:
Locations (1):
- Imelda General Hospital, Bonheiden, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hirten RP, Danieletto M, Sanchez-Mayor M, Whang JK, Lee KW, Landell K, Zweig M, Helmus D, Fuchs TJ, Fayad ZA, Nadkarni GN, Keefer L, Suarez-Farinas M, Sands BE. Physiological Data Collected From Wearable Devices Identify and Predict Inflammatory Bowel Disease Flares. Gastroenterology. 2025 May;168(5):939-951.e5. doi: 10.1053/j.gastro.2024.12.024. Epub 2025 Jan 16. PMID 39826619
- [Background] Ghosh S, Louis E, Beaugerie L, Bossuyt P, Bouguen G, Bourreille A, Ferrante M, Franchimont D, Frost K, Hebuterne X, Marshall JK, O'Shea C, Rosenfeld G, Williams C, Peyrin-Biroulet L. Development of the IBD Disk: A Visual Self-administered Tool for Assessing Disability in Inflammatory Bowel Diseases. Inflamm Bowel Dis. 2017 Mar;23(3):333-340. doi: 10.1097/MIB.0000000000001033. PMID 28146002
- [Background] Rowan C, Hirten R. The future of telemedicine and wearable technology in IBD. Curr Opin Gastroenterol. 2022 Jul 1;38(4):373-381. doi: 10.1097/MOG.0000000000000845. PMID 35762696
- [Background] Singh B, Chastin S, Miatke A, Curtis R, Dumuid D, Brinsley J, Ferguson T, Szeto K, Simpson C, Eglitis E, Willems I, Maher C. Real-World Accuracy of Wearable Activity Trackers for Detecting Medical Conditions: Systematic Review and Meta-Analysis. JMIR Mhealth Uhealth. 2024 Aug 30;12:e56972. doi: 10.2196/56972. PMID 39213525
- [Background] Louis S, Lembrechts N, Pouillon L. Towards a Greener IBD-Care: Let's INTERACT! United European Gastroenterol J. 2025 Mar;13(2):276-277. doi: 10.1002/ueg2.12728. Epub 2024 Dec 4. No abstract available. PMID 39632541
- [Background] Pouillon L, Hoefkens E, Verheyen V, Bronswijk M, Van Olmen A, Van Dessel S, Siborgs N, Bossuyt P. Letter to the Editor: Feasibility and Efficiency of an E-Health Preadmission Assessment System for Intravenous Therapy in Inflammatory Bowel Disease. Inflamm Bowel Dis. 2020 Jan 6;26(2):e11-e12. doi: 10.1093/ibd/izz304. No abstract available. PMID 31793628
- [Background] Bossuyt P, Hoefkens E, Pouillon L. Prime Time Was Yesterday for Patient-reported Outcomes in Daily Care of Patients With Inflammatory Bowel Diseases. Clin Gastroenterol Hepatol. 2018 Nov;16(11):1839. doi: 10.1016/j.cgh.2018.05.029. No abstract available. PMID 30343866
- [Background] Schoenfeld R, Nguyen GC, Bernstein CN. Integrated Care Models: Optimizing Adult Ambulatory Care in Inflammatory Bowel Disease. J Can Assoc Gastroenterol. 2018 Oct 15;3(1):44-53. doi: 10.1093/jcag/gwy060. eCollection 2020 Feb. PMID 34169226
- [Background] Turner D, Ricciuto A, Lewis A, D'Amico F, Dhaliwal J, Griffiths AM, Bettenworth D, Sandborn WJ, Sands BE, Reinisch W, Scholmerich J, Bemelman W, Danese S, Mary JY, Rubin D, Colombel JF, Peyrin-Biroulet L, Dotan I, Abreu MT, Dignass A; International Organization for the Study of IBD. STRIDE-II: An Update on the Selecting Therapeutic Targets in Inflammatory Bowel Disease (STRIDE) Initiative of the International Organization for the Study of IBD (IOIBD): Determining Therapeutic Goals for Treat-to-Target strategies in IBD. Gastroenterology. 2021 Apr;160(5):1570-1583. doi: 10.1053/j.gastro.2020.12.031. Epub 2021 Feb 19. PMID 33359090
- [Background] Magro F, Gionchetti P, Eliakim R, Ardizzone S, Armuzzi A, Barreiro-de Acosta M, Burisch J, Gecse KB, Hart AL, Hindryckx P, Langner C, Limdi JK, Pellino G, Zagorowicz E, Raine T, Harbord M, Rieder F; European Crohn's and Colitis Organisation [ECCO]. Third European Evidence-based Consensus on Diagnosis and Management of Ulcerative Colitis. Part 1: Definitions, Diagnosis, Extra-intestinal Manifestations, Pregnancy, Cancer Surveillance, Surgery, and Ileo-anal Pouch Disorders. J Crohns Colitis. 2017 Jun 1;11(6):649-670. doi: 10.1093/ecco-jcc/jjx008. No abstract available. PMID 28158501
- [Background] Harbord M, Eliakim R, Bettenworth D, Karmiris K, Katsanos K, Kopylov U, Kucharzik T, Molnar T, Raine T, Sebastian S, de Sousa HT, Dignass A, Carbonnel F; European Crohn's and Colitis Organisation [ECCO]. Third European Evidence-based Consensus on Diagnosis and Management of Ulcerative Colitis. Part 2: Current Management. J Crohns Colitis. 2017 Jul 1;11(7):769-784. doi: 10.1093/ecco-jcc/jjx009. No abstract available. PMID 28513805
- [Background] Adamina M, Minozzi S, Warusavitarne J, Buskens CJ, Chaparro M, Verstockt B, Kopylov U, Yanai H, Vavricka SR, Sigall-Boneh R, Sica GS, Reenaers C, Peros G, Papamichael K, Noor N, Moran GW, Maaser C, Luglio G, Kotze PG, Kobayashi T, Karmiris K, Kapizioni C, Iqbal N, Iacucci M, Holubar S, Hanzel J, Sabino JG, Gisbert JP, Fiorino G, Fidalgo C, Ellu P, El-Hussuna A, de Groof J, Czuber-Dochan W, Casanova MJ, Burisch J, Brown SR, Bislenghi G, Bettenworth D, Battat R, Atreya R, Allocca M, Agrawal M, Raine T, Gordon H, Myrelid P. ECCO Guidelines on Therapeutics in Crohn's Disease: Surgical Treatment. J Crohns Colitis. 2024 Oct 15;18(10):1556-1582. doi: 10.1093/ecco-jcc/jjae089. PMID 38878002
- [Background] Burisch J, Zhao M, Odes S, De Cruz P, Vermeire S, Bernstein CN, Kaplan GG, Duricova D, Greenberg D, Melberg HO, Watanabe M, Ahn HS, Targownik L, Pittet VEH, Annese V, Park KT, Katsanos KH, Hoivik ML, Krznaric Z, Chaparro M, Loftus EV Jr, Lakatos PL, Gisbert JP, Bemelman W, Moum B, Gearry RB, Kappelman MD, Hart A, Pierik MJ, Andrews JM, Ng SC, D'Inca R, Munkholm P. The cost of inflammatory bowel disease in high-income settings: a Lancet Gastroenterology & Hepatology Commission. Lancet Gastroenterol Hepatol. 2023 May;8(5):458-492. doi: 10.1016/S2468-1253(23)00003-1. Epub 2023 Mar 2. PMID 36871566
- [Background] Ng SC, Shi HY, Hamidi N, Underwood FE, Tang W, Benchimol EI, Panaccione R, Ghosh S, Wu JCY, Chan FKL, Sung JJY, Kaplan GG. Worldwide incidence and prevalence of inflammatory bowel disease in the 21st century: a systematic review of population-based studies. Lancet. 2017 Dec 23;390(10114):2769-2778. doi: 10.1016/S0140-6736(17)32448-0. Epub 2017 Oct 16. PMID 29050646
- [Background] Ungaro R, Mehandru S, Allen PB, Peyrin-Biroulet L, Colombel JF. Ulcerative colitis. Lancet. 2017 Apr 29;389(10080):1756-1770. doi: 10.1016/S0140-6736(16)32126-2. Epub 2016 Dec 1. PMID 27914657
- [Background] Torres J, Mehandru S, Colombel JF, Peyrin-Biroulet L. Crohn's disease. Lancet. 2017 Apr 29;389(10080):1741-1755. doi: 10.1016/S0140-6736(16)31711-1. Epub 2016 Dec 1. PMID 27914655